CLINICAL TRIAL: NCT07120087
Title: Evaluation of a Virtual Risk-reduction Intervention Among Women at Higher Than Average Risk of Breast Cancer in the European MyPeBS Screening Trial
Brief Title: Evaluation of an Online Intervention to Educate Women at High Risk of Breast Cancer on How to Help Reduce Their Risk.
Acronym: MyPREV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UC-BCG-2508
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Prevent and treat - breast cancer screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Other): intervention
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Virual Webinar and online personalised clinical visit

SUMMARY:
Breast cancer remains the most common cancer among women and a major cause of death despite advances in screening and treatment. Current screening programs are not personalized and are experiencing declining participation. A promising strategy for breast cancer control would be to implement risk-based prevention and early screening, targeting individuals at high risk of developing breast cancer, in order to improve chances of cure and reduce the need for more intensive treatments. The MyPeBS study was designed to assess whether personalized breast cancer screening (based on an individual's risk of developing breast cancer) is as effective as, or more effective than, current standard screening.

Lifestyle interventions involving changes in diet or physical activity, for example, have been shown to be effective in reducing the risk of developing breast cancer, whether low or high. The MyPeBS study evaluates personalized screening but offers limited information on breast cancer prevention. MyPREV is a project that aims to assess the feasibility and impact of a personalized online program on breast cancer risk reduction measures. This program is offered to women at high risk of developing breast cancer as part of the European MyPeBS screening study.

The main objective is to evaluate adherence to a personalized, online breast cancer prevention program focused on lifestyle and its acceptance among women at high or very high risk of developing cancer who participated in the MyPeBS study.

DETAILED DESCRIPTION:
MyPREV is a prospective interventional cohort study. The study is based on an online educational, medical, and motivational intervention (webinar and online personalized clinical visit) dedicated to promoting and implementing lifestyle-based breast cancer risk-reduction measures among women identified in the MyPeBS trial as being at high or very high risk of breast cancer based on Polygenic risk score (PRS) and clinical scores. In MyPeBS, 34.4% of the women in the risk-based arm were estimated to be at high (33.03%) or very high (1.37%) to develop a breast cancer within 5 years.

The study MyPREV plans to invite 3016 women (1821 in France and 1195 in Italy for the sites CPO and ISPRO). The expected participation rate is 50%, so around 1507 women (910 in France and 597 in Italy for the sites CPO and ISPRO). The intervention consist of a virtual webinar and an online personalized clinical visit where the personalized prevention plan will be created.

ELIGIBILITY:
Inclusion Criteria:

1. Female (whether born female or not)
2. Women aged 40 to 74 years (inclusive)
3. Women who have participated in, or are participating in the MyPeBS study and who fulfilled all the inclusion and non-inclusion criteria for the MyPeBS study.
4. Women able to express their non-opposition to participate in the intervention
5. Women who were assessed as being at high (≥≥1.67% - 5.9%) or very high (≥≥6%) risk of invasive breast cancer at 5 years in the MyPeBS study

Exclusion Criteria:

1. Women who developed a breast cancer during their follow-up in the MyPeBS study

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1508 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Acceptance | From start of the inclusion up to the end of inclusions
  To assess the acceptance of a full, targeted, online, educational and motivational intervention on breast cancer risk reduction measures among women who took part in MyPeBS and were identified to have a high or very high risk of breast cancer.

SECONDARY OUTCOMES:
Prevalence of risk reduction targets | From start of the inclusion up to the end of inclusions
  Assess the prevalence of breast cancer risk reduction targets (potentially modifiable factors) among women willing to participate
WCRF | At 3 months, 1 year
  Assess the participants' progress in modifying some of their behaviours according to the WCRF score at 3 months and 1 year
Strate-Trait Anxiety Inventory - State (STAI-S) | At baseline
  Evaluate patient characteristics (age, country, education level, professional occupation, Strate-Trait Anxiety Inventory [STAI] score at baseline in MyPeBS, level of breast cancer risk) associated with participation or non-participation in the proposed program and receipt of the proposed intervention
Subject knowledge and perception of knowledge | At baseline, 1 year
  Evaluate the knowledge and perception of knowledge regarding breast cancer risk and risk reduction measures with a specific questionnaire
Subject anxiety | At baseline, 1 year
  Subject anxiety will be evaluated using the State-Trait Anxiety Inventory (STAI) questionaire
Subject satisfaction | At baseline, 1 year
  Subject satisfaction will be measured using a specific questionnaire.
Levers and barriers for lifestyle modifications | At 1 year
  Evaluate the prevalence of predefined or self-assessed potential levers and barriers for lifestyle modifications

CONTACTS AND LOCATIONS:
Locations (2):
- Gustave Roussy, Villejuif, France
- AOU Città della Salute e della Scienza - CPO PiedmontSSD Epidemiologia e Screening, Torino, Italy

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported.
  A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.